CLINICAL TRIAL: NCT00595543
Title: Treatment of Acute Pseudophakic Cystoid Macular Edema: Bromfenac 0.09% Versus Diclofenac Sodium 0.1% Versus Ketorolac Tromethamine 0.5%
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bp Consulting, Inc (Network)
Responsible Party: David Rho, MD, Soll Eye Associates
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5349
Record Dates: First submitted 2008-01-07; First posted 2008-01-16 (Estimated); Last update posted 2009-03-19 (Estimated); Status verified 2009-03

CONDITIONS: Acute Pseudophakic Cystoid Macular Edema
MeSH Terms: interventions — bromfenac; Ketorolac; Diclofenac

ARMS (3):
- 1 (Active Comparator)
  Interventions: Drug: Bromfenac
- 2 (Active Comparator)
  Interventions: Drug: Ketorolac
- 3 (Active Comparator)
  Interventions: Drug: Diclofenac

INTERVENTIONS:
Drug: Bromfenac — 1 drop (in the eye) Instill one drop in the affected eye twice daily for three months
  Arms: 1
Drug: Ketorolac — 1 drop (in the eye) Instill one drop in the affected eye four times daily for three months
  Arms: 2
Drug: Diclofenac — 1 drop (in the eye) Instill one drop in the affected eye four times daily for three months
  Arms: 3

SUMMARY:
To compare bromfenac 0.09%, diclofenac sodium 0.1%, and ketorolac tromethamine 0.5% ophthalmic solutions for the treatment of acute pseudophakic CME after cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be diagnosed with acute pseudophakic CME within 12 months of cataract surgery
* Males and females 18 years and older
* Able to provide written informed consent

Exclusion Criteria:

* Complicated cataract surgery, particularly posterior capsule rupture and vitreous loss
* Pre-Existing macular pathology, including macular edema, macular scar, macular hole, or macular pucker
* History of Uveitis
* Ipsilateral intraocular surgery prior to cataract surgery
* CME greater than one year duration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Estimated)
Dates: Start 2008-01; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Acute Pseudophakic Cystoid Macular Edema | 5 months

SECONDARY OUTCOMES:
Visual Acuity | 5 months

CONTACTS AND LOCATIONS:
Overall Officials: David Rho, MD, Principal Investigator — Soll Eye Associates
Locations (1):
- Soll Eye Associates, Philadelphia, Pennsylvania, United States